CLINICAL TRIAL: NCT02273245
Title: Is a Pre-contrast Scan Necesary to Diagnose Acute Aortic Syndrome?
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 14/P/155
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Acute Aortic Syndrome
MeSH Terms: conditions — Acute Aortic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- thoracic aortgram CTs: A retrospective cohort assessment of thoracic aortogram CTs of male and female adult (age>18) patients presenting with symptoms of AAS.
  Interventions: Radiation: Thoracic aortogram CT

INTERVENTIONS:
Radiation: Thoracic aortogram CT — With and without contrast dye

SUMMARY:
Acute Aortic Syndrome (AAS) is a potentially life-threatening cause of sudden, severe chest pain. There are several possible underlying causes, which cannot be distinguished from one another at the bedside.

Current practice is to image this with two CT scans of the chest, one before injection of a contrast dye into the blood stream and then one after.

With the advancement of CT scanner technology, improvements in software interpretation and screen resolution, the investigators hypothesise that performing the contrast scan on its own is diagnostically equivalent to both the pre- and contrast scans

DETAILED DESCRIPTION:
AAS include: a tear in the wall of the main artery from the heart, bleeding directly into this wall, an ulcer in the wall, and excess dilatation and rupture of the main artery wall. These are also treated differently according to where they are in the length of the aorta. It is therefore important to identify precisely the subtype of AAS and its location to allow the clinician to manage the patient appropriately.

Current practice is to image this with two CT scans of the chest, one before injection of a contrast dye into the blood stream and then one after. The one before the contrast is used to determine if there is bleeding within the wall, which would show up as white on this scan. It is currently accepted that the contrast in the artery itself would hide the presence of bleeding within the wall. The other causes are seen primarily on the contrast scan only. Every patient proceeds from the pre-contrast scan to the contrast scan, unless there is a contraindication to the intravenous dye.

The investigators own database search has shown that radiologists protocol the scans according to their own preference and experience (i.e. some do both scans, others the contrast scan only). There is conflicting advice from international professional bodies as to whether to perform the non-contrast scan every time.

Some studies have shown that although the pre-contrast scan is sensitive to picking up bleeding within the wall, it adds nothing more over an increased radiation dose to the patient.

The investigators hypothesise that performing the contrast scan on its own is diagnostically equivalent to both the pre- and contrast scans to look for all 4 of these entities that make up AAS. The investigators also propose that not requiring the pre-contrast scan would have significant savings in patient radiation dose, scanner time, network resources and radiologist time.

ELIGIBILITY:
Inclusion Criteria:

* male and female adult (age>18) patients presenting with symptoms of AAS who had thoracic aortogram CTs.

Exclusion Criteria:

* age<18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective cohort assessment of thoracic aortogram CTs of male and female adult (age>18) patients presenting with symptoms of AAS.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Blinded review | 3 months
  2 experienced reporters are asked to blind view, in random order, either a contrast scan only, or a pair of pre- and post-contrast scans and report on an Excel spreadsheet.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Roobottom, MBChB FRCP, Study Director — Plymouth Hospital NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom